CLINICAL TRIAL: NCT05063968
Title: A Phase I Clinical Trial to Evaluate the Safety Tolerability Pharmacokinetics (PK) of XZP-6019 Tablets Following Single- and Multiple-ascending Doses (SAD/MAD) and Food Effects in Healthy Subjects
Brief Title: A Clinical Trial of XZP-6019 Tablets in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6019-CPK-1001
Record Dates: First submitted 2021-09-21; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A - Single Ascending Dose (SAD) phase: Experimental (Experimental)
  Interventions: Drug: XZP-6019 tablet
- Part A - Single Ascending Dose (SAD) phase:Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B - Food Effect (FE) phase: Experimental 1 (Experimental)
  Interventions: Drug: XZP-6019 tablet
- Part B - Food Effect (FE) phase: Experimental 2 (Experimental)
  Interventions: Drug: XZP-6019 tablet
- Part C - multiple ascending dose (MAD) phase: Experimental (Experimental)
  Interventions: Drug: XZP-6019 tablet
- Part C - multiple ascending dose (MAD) phase:Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XZP-6019 tablet — Tablet is administered orally once on Day 1 and Day 9, respectively
  Arms: Part A - Single Ascending Dose (SAD) phase: Experimental
Drug: Placebo — Tablet is administered orally once on Day 1 and Day 9, respectively
  Arms: Part A - Single Ascending Dose (SAD) phase:Placebo
Drug: XZP-6019 tablet — Tablet is administered fasted orally once on Day 1
  Arms: Part B - Food Effect (FE) phase: Experimental 1
Drug: XZP-6019 tablet — Tablet is administered after a high-fat meal orally once on Day 9
  Arms: Part B - Food Effect (FE) phase: Experimental 2
Drug: XZP-6019 tablet — Tablet is administered orally once daily for 14 Days continuously
  Arms: Part C - multiple ascending dose (MAD) phase: Experimental
Drug: Placebo — Tablet is administered orally once daily for 14 Days continuously
  Arms: Part C - multiple ascending dose (MAD) phase:Placebo

SUMMARY:
This study will consist of 3 parts: Part A - Single Ascending Dose (SAD) phase, Part B - Food Effect (FE) phase, and Part C - multiple ascending dose (MAD) phase.

DETAILED DESCRIPTION:
Part A and Part C studies were designed as single-center, randomized, double-blind, placebo-controlled, dose-escalation trials to assess the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles of single and multiple oral doses of XZP-6019 tablets in healthy adult subjects. Part B is a single-center, randomized, open label, 2×2 crossover design to assess the food effects on PK of a single oral dose of XZP-6019 tablets in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria will be enrolled in this study.

  1. Healthy adult males or females aged 18 to 45 years (including 18 and 45 years old).
  2. Body weight ≥ 50 kg for males and ≥ 45 kg for female; body mass index (BMI) in the range of 19.0-26.0 kg/m2 for the non-obese cohort and in the range of 28.1 -35.0 kg/m2 for the obese cohort (including the boundary value, BMI=weight/height2).
  3. No plans for childbearing or donating sperm/egg within the latest 6 months, and willing to use effective contraception within 6 months after the end of dosing
  4. No clinically significant findings in vital signs, physical examination, laboratory tests, or ECG or Lung CT for Low-dose.
  5. Subjects understand and comply with the study procedures, voluntarily participate, and sign an Informed Consent Form.

Exclusion Criteria:

* Subjects meeting any of the following criteria will not be enrolled in this study:

  1. With history or presence of clinically significant abnormalities, e.g.: significant abnormality or disease of endocrine, gastrointestinal, cardiovascular, hematologic, hepatic, immunologic, renal, respiratory, genitourinary or major neurological (including stroke and chronic epilepsy) or patients with psychosomatic disorders
  2. History of clinically significant ECG abnormalities or family history of long QT syndrome (grandparents, parents and siblings), or

     Any of the following was regarded as a criterion for exclusion:
     1. Confirmation of QTcF ≥ 450 ms by repeated measurements;
     2. Confirmation of QRS duration > 120 ms by repeated measurements;
     3. Confirmation of PR interval > 200 ms by repeated measurements;
     4. Findings that make QTc measurement difficult or QTc data difficult to interpret;
     5. History of other risk factors for Torsades de Pointes tachycardia (e.g., heart failure, hypokalemia, family history of long QT syndrome);
     6. Presence of uncorrected hypokalemia or hypomagnesemia.
  3. Subjects with a known or suspected history of allergy to the test drug or its excipient components, or a history of clinically significant severe allergy (e.g., food, drug, latex allergy), or a history of atopic allergic disease (asthma, urticaria, eczematous dermatitis)
  4. History of dysphagia or any gastrointestinal disorder affecting drug absorption at screening, including history of frequent nausea or vomiting of any etiology, history of irregular gastrointestinal motility such as habitual diarrhea, constipation or pre-irritable bowel syndrome, or history of major gastrointestinal surgery (e.g., gastrectomy, gastrointestinal anastomosis, bowel resection, gastric bypass, gastric division, or gastric banding)
  5. History of pancreatic injury or pancreatitis at screening, or significantly elevated blood amylase (> 1.5 ULN)
  6. History of urinary tract obstruction or presence of urinary voiding difficulties at screening.
  7. History of cancer (malignancy) at the time of screening.
  8. Positive test results for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or syphilis antibody
  9. History of significant drug abuse within 12 months prior to screening or positive urinary drug test at screening
  10. Regular alcohol consumption within 3 months prior to screening, consuming more than 3 alcoholic drinks per day (one drink is approximately equal to: beer 354 mL/12 oz, wine 118 mL/4 oz, or distilled spirits 29.5 mL/1 oz), or evidence of alcohol abuse and excessive consumption as evidenced by alcohol breath test at screening (subjects consuming 4 alcoholic drinks per day may be enrolled at the discretion of the investigator).
  11. History of smoking within 3 months prior to screening, or a positive urinary nicotine test at screening, or who cannot give up smoking throughout the study period
  12. Excessive daily intake of coffee, tea, cola, energy drinks, or other caffeinated beverages within 3 months prior to screening, with excess defined as more than 6 servings (one serving is approximately equal to 120 mg of caffeine).
  13. Major surgery, or donation or loss of blood over 400 mL within 3 months prior to administration.
  14. Participation in other clinical trials and treatment with investigational product within 3 months prior to administration.
  15. Take any prescription, over-the-counter, health product, herbal or proprietary Chinese medicine within 4 weeks prior to administration (or less than 5 half-lives of the drug administration from the start of the trial).
  16. Women who are pregnant or breastfeeding, or of childbearing potential who are not using effective non-hormonal contraception (intrauterine device (IUD), barrier method with spermicide, or surgical sterilization, etc.) or are unwilling to continue using these methods during the trial until 6 months after discontinuation; men of childbearing potential who are unwilling to use physical methods of contraception during the trial until 6 months after discontinuation.
  17. At the time of screening, Systolic blood pressure ≥ 140 mmHg or < 90 mmHg, and/or diastolic blood pressure ≥ 90 mmHg or < 50 mmHg.
  18. At the time of screening, Heart rate < 50 or > 100 beats/min.
  19. Glomerular filtration rate (eGFR) < 90 ml/min/1.73m2 was estimated at screening according to the Chronic Kidney Disease Epidemic (CKD-EPI) formula (see Annex 1 for calculation formula).
  20. At screening, the liver function tests showed any measure of aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) or total bilirubin is > upper limit of normal (ULN) in non-obesity cohorts; liver function tests of obese group showed AST, ALT or ALP is > 1.5 ULN, or total bilirubin is > ULN in obesity cohort.
  21. Fasting triglycerides > 2.3mmol/L at the time of screening.
  22. Fasting glucose > 5.6 mmol/L in the non-obese cohort and > 6.1 mmol/L or glycosylated hemoglobin (HbA1c) ≥ 6.5% in the obese group at screening.
  23. Those who could not tolerate blood sample collection.
  24. Subjects who are deemed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Prior to dosing, 0.25,0.5,1,2,3,4,6,8,12,24,36,48,72 hours post dose.
Tmax | Prior to dosing, 0.25,0.5,1,2,3,4,6,8,12,24,36,48,72 hours post dose.
AUC0-t | Prior to dosing, 0.25,0.5,1,2,3,4,6,8,12,24,36,48,72 hours post dose.
AUC0-inf | Prior to dosing, 0.25,0.5,1,2,3,4,6,8,12,24,36,48,72 hours post dose.
T1/2 | Prior to dosing, 0.25,0.5,1,2,3,4,6,8,12,24,36,48,72 hours post dose.
CL/F | Prior to dosing, 0.25,0.5,1,2,3,4,6,8,12,24,36,48,72 hours post dose.
Vz/F | Prior to dosing, 0.25,0.5,1,2,3,4,6,8,12,24,36,48,72 hours post dose.
Subject incidence of adverse events for XZP-6019 versus placebo | Part A: From signing Informed consent form to Day 16; Part B: From signing Informed consent form to Day 16; Part C: From signing Informed consent form to Day 42.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Dong, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No